CLINICAL TRIAL: NCT06958952
Title: Evaluating the Efficacy of "Digestive Aid" in Functional Dyspepsia: A Randomized Double Blind Control Trial
Brief Title: Evaluating the Efficacy of "Digestive Aid" in Functional Dyspepsia
Acronym: Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Darman Yab Darou Co. (Unknown)
Responsible Party: Principal Investigator, Raika Jamali, MD, Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1403-4-101-75896; 1403-4-101-75896 (Other: Tehran University of Medical Sciences)
Record Dates: First submitted 2025-03-07; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Dyspepsia Chronic
Keywords: Efficacy; Clinical trial; Functional Dyspepsia; questionnaire; Digestive Aid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digestive Aid (Experimental): Treatment with Digestive Aid
  Interventions: Dietary Supplement: Digestive Aid
- Placebo (Placebo Comparator): Treatment with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Digestive Aid — one tablet daily for one month
  Arms: Digestive Aid
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Functional Dyspepsia (FD) is diagnosed in the presence of bothersome epigastric pain or burning, early satiation and/or postprandial fullness of greater than 8 weeks duration, in the absence of alarm signs. Alarm signs include weight loss, gastrointestinal bleeding, anemia, dysphagia, and family history of upper gastrointestinal malignancies. FD is a common gastrointestinal complaint. It's prevalence in Iranian population is reported to be from 2.2% to 29.9% (1). FD should be introduced as a disorder of gut-brain interaction (DGBI), together with a simple account of the gut-brain axis and how this is impacted by diet, stress, cognitive, behavioral and emotional responses to symptoms and post-infective changes. Histamine-2-receptor antagonists, proton pump inhibitors, and prokinetics are introduced as the first line classic treatment in FD. (2) Tricyclic antidepressants (TCAs) used as gut-brain neuromodulators are an efficacious second-line treatment for FD. (2) Antipsychotics, such as sulpiride 100 mg four times a day or levosulpiride 25 mg three times a day, may be efficacious as a second-line treatment for FD. Tandospirone, Pregabalin, Mirtazapine are among the suggested second line pharmachological therapy. (2) FD expresses a spectrum of various upper gastrointestinal complaints. Epigastric pain, retrosternal pain, regurgitation, nausea, vomiting, belching, dysphagia, and early satiety are among the most frequent symptoms. Therefore, a combination of medications might be needed to alleviate the patients' discomfort. The pharmaceutics have proposed the package of medications to increase the patient compliance. "Digestive Aid" is a cocktail that contains Marshmallow, Ginger, Gentian, Fennel, Peppermint, and Anise oil. It is widely used by physicians to control dyspeptic symptoms. There are studies on human and animals that showed the efficacy of mentioned herbal supplements on dyspepsia. To the best of our knowledge there is no study about the efficacy of "Digestive Aid" in the dyspeptic patients. This trial is conducted to evaluate the efficacy of mentioned product in alleviating the symptoms in FD in a sample of the Iranian patients.

DETAILED DESCRIPTION:
This double blind placebo-control clinical trial is performed in dyspeptic patients referred to the gastroenterology clinic in Sina Hospital. Neither the participants nor the researcher knows which treatment or intervention are provided until the end of trial. The new onset dyspeptic patients that are older than 18 years of age will be included in the project. The gastroenterologist diagnose FD after taking the complete medical history, physical examination, laboratory investigations and performing upper gastrointestinal endoscopy. Participants with co-morbidities (known GI diseases), taking medications, those with abnormal gastrointestinal findings in physical examination and para-clinical investigations will be excluded from the research. FD will be diagnosed based on the Rome 4 criteria.

Participants will fill out an informed written consent prior to the enrollment. The trial has two arms. The patients in case group receive the film-coated "Digestive Aid" product once daily for 2 months. The control group takes the placebo for the same duration. Both products are manufactured by Darman Yab Darou Incorporation, Tehran, Iran. The caregiver who gives the medication to the participants is blind to the type of capsules. Block Randomization will be used to assign the participants to intervention or placebo group considering their age and gender.

The efficacy of medication on the severity of symptom is evaluated by the valid Persian version of the "Leeds dyspepsia questionnaire" (LDQ).(3) This questionnaire evaluates 8 dyspeptic complaints. Epigastric pain, retrosternal pain, regurgitation, nausea, vomiting, belching, dysphagia, and early satiety are the key elements that are evaluated in this questionnaire. The severity of symptoms are graded from 0 to 8. The sum of scores in all 8 items of the questionnaire represents the patients' total score. The Primary outcome measure is defining the changes of dyspeptic symptoms from baseline to the end of treatment.

A statistical power analysis is used to calculate the sample size. Considering the two-sided significant level (α) of 0.05 and the power of 90% (β = 0.1), a total sample size of 46 patients is determined to detect one percent inter-group difference in LDQ score. (For detailed information, please refer to http://hedwig.mgh.harvard.edu/sample_size/js/js_parallel_quant.html). To allow for a 5% possible dropout rate, 50 patients will be recruited in the trial.

Analysis of covariance (ANCOVA) will be applied for comparing treatment groups regarding the changes of variables during the study. All statistical analyses will be performed using SPSS version 17 (SPSS, Chicago, IL, The USA). The probability of the difference between the dependent and independent variables is considered significant if a two-tailed P value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The new onset dyspeptic patients

Exclusion Criteria:

* Participants with co-morbidities (known GI diseases)
* Taking medications,
* Those with abnormal gastrointestinal findings in physical examination and para-clinical investigations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Functional Dyspepsia | One month
  Functional Dyspepsia evaluation based on the Leeds Dyspepsia Questionnaire (LDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Professor
Locations (1):
- Sina Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
All the data

REFERENCES:
- [Result] Amini E, Keshteli AH, Jazi MS, Jahangiri P, Adibi P. Dyspepsia in Iran: SEPAHAN Systematic Review No. 3. Int J Prev Med. 2012 Mar;3(Suppl 1):S18-25. PMID 22826763
- [Result] Narendren A, Boddupalli S, Segal JP. British Society of Gastroenterology guidelines on the management of functional dyspepsia. Frontline Gastroenterol. 2023 Oct 11;15(1):70-73. doi: 10.1136/flgastro-2023-102508. eCollection 2024 Jan. PMID 38487566
- [Result] Batebi S, Masjedi Arani A, Jafari M, Sadeghi A, Saberi Isfeedvajani M, Davazdah Emami MH. Validity and Reliability of the Persian Version of Leeds Dyspepsia Questionnaire. Galen Med J. 2019 Dec 31;8:e1609. doi: 10.31661/gmj.v8i0.1609. eCollection 2019. PMID 34466536